CLINICAL TRIAL: NCT05506332
Title: ABT-199 (Venetoclax) and Purine Analogues as Novel Oral Drug Combination for Treatment of Relapsed/Refractory Acute Myeloid Leukemia: the ApoAML Trial
Brief Title: Treatment With ABT-199 (Venetoclax) and Purine Analogues in Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2282; 2021-006473-35 (EudraCT Number)
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Mercaptopurine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax and 6-mercaptopurine (Experimental): Single arm study with venetoclax and 6-mercaptopurine administered in two to six cycles of 28 days. Venetoclax is given at a dosage of 600mg with dose reduction in case of interaction with a moderate or strong CYP3A4 inhibitor. 6-mercaptopurine is given at a dosage of 100mg.
  Interventions: Drug: Venetoclax; Drug: 6-mercaptopurine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax and 6-mercaptopurine
Drug: 6-mercaptopurine — Venetoclax and 6-mercaptopurine

SUMMARY:
Non-commercial, open-label interventional phase Ib study to assess the effectivity of the combination of venetoclax and 6-mercaptopurine in patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
Non-commercial, open-label interventional phase Ib study. The aim of the study is to assess the effectivity of the combination of venetoclax and 6-mercaptopurine in patients with relapsed or refractory AML.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory AML
* Relapsed after or refractory to at least one cycle of intensive chemotherapy (combination of ara-c/anthracyclin) or four cycles of HMA (hypomethylating agents)
* Adult AML aged >/= 18 years
* WHO performance status: grade 0-2 at the time of enrollment
* ABT-199 (venetoclax) and PA-naïve. Patient may be prior exposed but not refractory to venetoclax. In case of previous therapy with venetoclax inclusion is only possible after discussion with the PI.

Exclusion Criteria:

* Participation in any other interventional clinical trial during the study period
* Active presence (or known history of) central nervous system disease
* History or concomitant presence of any other malignancy, except for non-melanoma skin cancer, carcinoma in situ of the cervix, any other effectively treated malignancy that has been in remission for >5 years or that is highly likely to be cured at the time of enrollment.
* Active HIV, hepatitis B or hepatitis C infection
* Use of any antitumoral agent within less than 5 times the half-life of the agent prior to the screening bone marrow examination. After the screening bone marrow examination, the use of cytoreductive treatment prior to the initiation of venetoclax is permitted in order to lower the WBC-count to <25 000/µl (e.g. hydroxyurea).
* Medical conditions requiring chronic therapy of moderate or strong CYP3A4 inducers without alternative
* Patients with known hypersensitivity to the active substance or to any of the excipients
* Pregnant or breastfeeding woman
* Active uncontrolled systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response | at 2 months
  Objective response rate
Clinical response | at 6 months
  Objective response rate
Clinical response | at 2 years
  Objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Anguille, Prof. Dr., Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Edegem, Antwerp
  - AZ Delta, Roeselare, West Vlaanderen

IPD SHARING:
Plan to Share IPD: No